CLINICAL TRIAL: NCT03027258
Title: Point-of-Delivery Prenatal Test Results Through mHealth to Improve Birth Outcome
Acronym: mHealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Echezona Ezeanolue, Professor of Public Health and Pediatrics, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 820085-3; R21TW010252-01 (NIH)
Record Dates: First submitted 2017-01-06; First posted 2017-01-23 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: HIV; Sickle Cell Disease; Hepatitis B
Keywords: Mobile health technology
MeSH Terms: conditions — Anemia, Sickle Cell; Hepatitis B | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): mHealth intervention
  Interventions: Other: mHealth

INTERVENTIONS:
Other: mHealth — HBI participants who consent will be enrolled in this study and will have data collected from their community screening stored in a secure, web-based database. The stored data will be encrypted into a Quick Response code embedded in a "smart card." A unique identification number and participant's blood group type will be on the outside of the card. There will be no names or any other identifiers. Each participating center will identify a dedicated delivery room staff that will be trained to read the contents of the card using the cell phone application as well as enter new data in the participant's profile. When a participant presents at delivery without the card, information can still be obtained from the secure, web-based database and confirmed using the participant's name, date of birth and cell phone number. This information is provided to the clinician to guide management of the infant.

SUMMARY:
The investigators propose to adopt sustainable community networks (in this case churches) to implement an integrated community-based screening that incorporates mobile health technology (mHealth) to make prenatal test results available at the point-of-delivery to guide medical management.

DETAILED DESCRIPTION:
The investigators will develop and test the feasibility, acceptability, and usability of a mobile health platform that captures results for HIV, Hepatitis B virus (HBV) and sickle cell genotype obtained from participants during the Healthy Beginning Initiative (HBI) program; store data in a secure, web-based database; encrypt data on a "smart card" which is given to participants, and make these data available at the point-of-delivery using a cell-phone application to read the "smart card". Data on the web-based database can also be accessed directly using the cell phone application. Evidence exists that when clinician have maternal records available at the point of delivery, they are more likely to initiate antiretroviral prophylaxis for HIV-exposed infants, administer the first dose of hepatitis B vaccine with 24 hours for infants born to women who have positive hepatitis B surface antigen and screen infants born to mothers with sickle cell trait to allow early identification and initiation of penicillin prophylaxis for infants who have sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women; 18 years or older enrolled in the Healthy Beginning Initiative
* One of the three conditions - HIV, Hepatitis B, and Sickle cell trait/disease

Exclusion Criteria:

* Those who do not accept to have their information uploaded on the secure database

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Reach | 6 months
  Reach will be calculated as: the proportion of enrolled pregnant women relative to eligible pregnant women in the study catchment area.
Effectiveness | 6 months
  Effectiveness will be determined by assessing the impact of the mHealth platform on key outcomes such as screening for HIV, HBV, and sickle cell genotype, and health care utilizations for follow up visits. This will be measured by calculating the percentage of pregnant women that used the "smart card" at the point-of-delivery.
Adoption | 6 months
  Adoption rates will be calculated using the proportion of interested health care settings to the total number eligible for participation.
Acceptability | 6 months
  The proportion of enrolled pregnant women who accept to use the smart card for their health care services

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Caritas Foundation, Makurdi, Benue State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezeanolue EE, Obiefune MC, Yang W, Obaro SK, Ezeanolue CO, Ogedegbe GG. Comparative effectiveness of congregation- versus clinic-based approach to prevention of mother-to-child HIV transmission: study protocol for a cluster randomized controlled trial. Implement Sci. 2013 Jun 8;8:62. doi: 10.1186/1748-5908-8-62. PMID 23758933
- [Derived] Gbadamosi SO, Eze C, Olawepo JO, Iwelunmor J, Sarpong DF, Ogidi AG, Patel D, Oko JO, Onoka C, Ezeanolue EE. A Patient-Held Smartcard With a Unique Identifier and an mHealth Platform to Improve the Availability of Prenatal Test Results in Rural Nigeria: Demonstration Study. J Med Internet Res. 2018 Jan 15;20(1):e18. doi: 10.2196/jmir.8716. PMID 29335234
- [Derived] Ezeanolue EE, Gbadamosi SO, Olawepo JO, Iwelunmor J, Sarpong D, Eze C, Ogidi A, Patel D, Onoka C. An mHealth Framework to Improve Birth Outcomes in Benue State, Nigeria: A Study Protocol. JMIR Res Protoc. 2017 May 26;6(5):e100. doi: 10.2196/resprot.7743. PMID 28550003